CLINICAL TRIAL: NCT01024361
Title: CPAP Application at Delivery Room at Very Low Birth Weight Infants
Brief Title: Cpap at Delivery Room for Preterm Infants
Acronym: CPAP-DR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Francisco Eulogio Martinez/ Professor Titular, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 120789; FAPESP 06/61388-2 (Other Grant/Funding Number: FAPESP 06/61388-2)
Record Dates: First submitted 2009-11-27; First posted 2009-12-02 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Mechanical Ventilation; Retinal Disease; Death; Respiratory Tract Disease
Keywords: Preterm infants; Nasal CPAP; Delivery room; Newborn
MeSH Terms: conditions — Retinal Diseases; Death; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Routine (No Intervention): Routine protocol of the service
- CPAP-DR (Experimental): Infants randomized to this arm will have nasal CPAP installation at delivery room before the 15th minute of life
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP of 5 cm water pressure will be applied within 15 minutes after birth by Neopuff
  Other Names: Neopuff
  Arms: CPAP-DR

SUMMARY:
The objective of the study is to determine if CPAP applied within less than 15 min of life in the DR reduces the necessity of mechanical ventilation and surfactant during the first 5 days of life.

DETAILED DESCRIPTION:
A multicenter prospective cohort of inborn preterm infants, born at 8 public university NICU in Brazil, with birthweight 1000-1499 g, without malformations, not intubated at 15 minutes of life. Preterm infants will be randomly assigned at birth to an early treatment group (DR-CPAP), in which CPAP of 5 cm water pressure is applied within 15 minutes after birth by Neopuff, or to a routine group (RG), in which CPAP is applied when indicated by the assistant physician. After transfer to the NICU, nasal CPAP will be maintained with Hudson prongs

ELIGIBILITY:
Inclusion Criteria:Inborn.

* Birth weight 1000g to 1500g
* No major malformations

Exclusion Criteria:

* Necessity of intubation
* Maternal decision

Ages: 1 Minute to 15 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Necessity of mechanical ventilation and surfactant during the first 5 days of life | 5 days

SECONDARY OUTCOMES:
Maternal and infant characteristics associated with CPAP failure during the first 15 minutes of life | 15 minutes
Incidence of pneumothorax, interstitial emphysema, ductus arteriosus, peri- intra-ventricular hemorrhage, sepsis, necrotizing enterocolitis | 30 days
Oxygen use | 28 days
Oxygen use | 56 days
Oxygen use | 36 weeks of corrected age
Retinopathies of prematurity | Hospital stay
Death during hospitalization | Hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Francisco E Martinez, MD, Principal Investigator — University of sao Paulo at Ribeirão Preto